CLINICAL TRIAL: NCT06286033
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AG-181 in Healthy Participants
Brief Title: Single and Multiple Ascending Dose Study and Food Effect Study for AG181
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG181-C-001
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: There are 3 parts in this study. Part 1 and 2 follows a sequential design. Part 3 is a food effect study with a 2x2 crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Single Ascending Dose (SAD) (Experimental): Participants will receive a range of doses of AG-181 or placebo, orally, once on Day 1. AG-181 will be given under fasted conditions.
  Interventions: Drug: AG-181; Drug: Placebo
- Part 2: Multiple Ascending Dose (MAD) (Experimental): Participants will receive a range of doses of AG-181 or placebo twice daily (BID) for 13 days and a single dose on Day 14 under fasted conditions.
  Interventions: Drug: AG-181; Drug: Placebo
- Part 3: Food Effect - Sequence 1: AB (Experimental): Participants will receive single oral dose of AG-181 on Day 1 of Period 1 under fasted condition (A) followed by single oral dose of AG-181 on Day 1 of Period 2 under fed (high fat meal) condition (B). Each period will be separated by a washout period of 1 week.
  Interventions: Drug: AG-181
- Part 3: Food Effect - Sequence 2: BA (Experimental): Participants will receive a single oral dose of AG-181 on Day 1 of Period 1 under fed (high fat meal) condition (B) followed by single oral dose of AG-181 on Day 1 of Period 2 under fasted condition (A). Each period will be separated by a washout period of 1 week.
  Interventions: Drug: AG-181

INTERVENTIONS:
Drug: AG-181 — AG-181 tablets
Drug: Placebo — AG-181 matched-placebo tablets
  Arms: Part 1: Single Ascending Dose (SAD); Part 2: Multiple Ascending Dose (MAD)

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of AG-181 in healthy participants after oral administration of single ascending dose (SAD) of AG-181 in Part 1 and multiple ascending dose (MAD) in Part 2 along with the effect of food on the pharmacokinetics (PK) of single oral doses of AG-181 in healthy participants in Part 3.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study, give written informed consent, and comply with the study restrictions.
* Body mass index in the range of 18.0 to 30.0 kilograms per square meter (kg/m^2).
* Weight ≥ 50 kilograms (kg) at screening.
* Healthy status as defined by the absence of evidence of any clinically significant, in the opinion of the Investigator, active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, serology, and urinalysis.
* Ability and willingness to refrain from alcohol-, caffeine-, and methylxanthine-containing beverages or food (e.g., coffee, tea, cola, chocolate, energy drinks) from 72 hours (3 days) before administration of the first dose of study drug through follow-up.
* All values for hematology and clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations, as judged by the Investigator.
* For women of child bearing potential (WOCBP)*, have a negative serum pregnancy test at Screening and during admission to the clinic.

  a. *WOCBP are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion; or who have not been naturally postmenopausal. WOCBP must use an acceptable method of contraception from Screening and until 14 days or 5 half-lives of AG-181, whichever is longer, after last dose of AG-181. WOCBP using hormonal contraception as a highly effective form of contraception must also use an acceptable barrier method.
* Male participants with female partners of childbearing potential must use a condom during treatment and for 14 days or 5 half-lives of AG-181, whichever is longer, after last dose of AG-181.
* Male participants must agree not to donate sperm during the study and for 14 days or 5 half-lives of AG-181, whichever is longer, after the last dose of study drug.
* Postmenopausal women are women who have not menstruated at all for at least the 12 months before providing informed consent and who have an elevated follicle-stimulating hormone (FSH) level indicative of menopause during screening.
* Participants must have discontinued use of prescription drugs (including topical skin preparations other than nonsteroidal/nonantibiotic nonprescription moisturizers) within 2 weeks or 5 half-lives (whichever is longer) of the first dose of study drug, and over-the-counter (OTC) medication (excluding routine vitamins) within 7 days of the first dose of study drug, unless agreed as not clinically relevant by the Investigator and Medical Monitor (or designee).

Exclusion Criteria:

* Women who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 14 days or 5 half-lives of AG-181, whichever is longer, after last dose of study drug.
* Males with female partners who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 14 days or 5 half-lives of AG-181, whichever is longer, after last dose of study drug.
* Prior exposure to AG-181.
* Use of any investigational drug or device within 30 days before administration of the first dose of study drug.
* Any disease which, in the opinion of the Investigator, poses an unacceptable risk to the participants.
* Clinically significant history of, including treatment within an Emergency Department for, any drug sensitivity, drug allergy, or food allergy, as determined by the Investigator (such as anaphylaxis, hepatotoxicity, or treatment with steroids or epinephrine).
* Creatinine clearance <90 milliliters per minute (mL/min) (by Cockcroft-Gault formula) at screening.
* Aspartate aminotransferase >upper limit of normal (ULN) or alanine aminotransferase >ULN at screening.
* Use of tobacco or nicotine products in the 48 hours (2 days) prior to administration of the first dose of study drug.
* Strenuous activity, sunbathing, and contact sports within 48 hours (2 days) prior to administration of the first dose of study drug.
* History of donation of more than 450 milliliters (mL) of blood within 60 days prior to administration of the first dose of study drug.
* Plasma or platelet donation within 7 days prior to administration of the first dose of study drug.
* History within the 12 months before Screening of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink=12 ounce (oz) beer, 5 oz wine, and 1.5 oz spirits). Alcohol consumption will be prohibited 72 hours prior to administration of the first dose of study drug and until discharge.
* Positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or anti-human immunodeficiency virus (HIV) 1 and 2 antibodies at screening.
* Consumption of any nutrients known to modulate cytochrome P450 (CYP450) enzymes activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, or Seville [blood] orange products) within 14 days prior to administration of the first dose of study drug.
* Positive alcohol or drug screen (cannabinoids, amphetamines, methamphetamines, 3,4-methylenedioxy-N-methylamphetamine [ecstasy], opiates, methadone, oxycodone, phencyclidine, cocaine, cotinine, benzodiazepines, and barbiturates) at screening or admission to the clinical facility.
* Prolonged heart rate-corrected QT interval (QTc) [heart rate-corrected QT interval by Fridericia's formula (QTcF) >450 milliseconds (msec)] during screening and prior to first dose of study drug.
* History of long-QT syndrome, torsade de pointes, or any risk factors for torsades de pointes in the opinion of the investigator.
* A history in any family member of any of the following: sudden cardiac death, unexplained death, long-QT syndrome, or death from a primary dysrhythmia potentially associated with QT prolongation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
SAD: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) by Type, Severity, and Relationship to Study Drug | Up to Day 7
MAD: Number of Participants with AEs and SAEs by Type, Severity, and Relationship to Study Drug | Up to Day 26
Food Effect: Maximum Observed Plasma Concentration (Cmax) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
Food Effect: Area Under the Concentration-time Curve up to the Last Quantifiable Concentration (AUC0-last) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
Food Effect: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
Food Effect: Time to Reach Maximum Observed Concentration (tmax) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
Food Effect: Terminal Elimination Rate Constant (Kel) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
Food Effect: Terminal Elimination Half-Life (t1/2) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
Food Effect: Apparent Oral Clearance (CL/F) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
Food Effect: Apparent Volume of Distribution at Terminal Phase (Vz/F) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4

SECONDARY OUTCOMES:
SAD: Maximum Observed Plasma Concentration (Cmax) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
SAD: Time to Reach Maximum Observed Concentration (tmax) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
SAD: Terminal Elimination Rate Constant (Kel) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
SAD: Terminal Elimination Half-Life (t1/2) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
SAD: Area Under the Concentration-time Curves (AUCs) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
SAD: Apparent Oral Clearance (CL/F) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
SAD: Apparent Volume of Distribution at Terminal Phase (Vz/F) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 4
SAD: Renal Clearance (CLR) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 3
SAD: Total Percent of AG-181 Dose Excreted Unchanged in Urine (Fet%) | Predose and multiple time points postdose from Day 1 to Day 3
SAD: Percent of AG-181 Dose Excreted Unchanged in Urine Between Time 1 and Time 2 (Fet1-t2%) | Predose and multiple time points postdose from Day 1 to Day 3
SAD: Cumulative Amount of AG-181 Drug Excreted in Urine (Ae0-t) | Predose and multiple time points postdose from Day 1 to Day 3
SAD: Amount of AG-181 Drug Excreted in Urine Between Time 1 and Time 2 (Aet1-t2) | Predose and multiple time points postdose from Day 1 to Day 3
MAD: Maximum Observed Plasma Concentration (Cmax) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 17
MAD: Time to Reach Maximum Observed Concentration (tmax) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 17
MAD: Terminal Elimination Rate Constant (Kel) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 17
MAD: Terminal Elimination Half-Life (t1/2) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 17
MAD: Area Under the Concentration-time Curve (AUC) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 17
MAD: Apparent Oral Clearance (CL/F) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 17
MAD: Apparent Volume of Distribution at Terminal Phase (Vz/F) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 17
MAD: Time to Maximum Observed Plasma Concentration at Steady State (Cmax_ss) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 17
MAD: Accumulation Ratio for Cmax (RA_Cmax) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 14
MAD: Accumulation Ratio for Area Under the Concentration-time Curve (RA_AUC) of AG-181 | Predose and multiple time points postdose from Day 1 to Day 14
Food Effect: Number of Participants with AEs and SAEs by Type, Severity, and Relationship to Study Drug | Up to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- ICON 1255 East 3900 South, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No